CLINICAL TRIAL: NCT05081752
Title: Comparison of no Fixation vs. Stent Suturing vs. OTSC Stentfix in Preventing Esophageal Stent Migration in Esophageal Strictures
Brief Title: Preventing Esophageal Stent Migration in Esophageal Strictures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruiting and lack of interest from care providers.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-01901
Record Dates: First submitted 2021-09-30; First posted 2021-10-18 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Stent Migration

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects will be blinded as to which study arm they are in, in order to avoid any bias they may have.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- No fixation (No Intervention)
- Stent Suturing (Active Comparator)
  Interventions: Procedure: Stent Suturing / Endoscopic Clips
- OTSC Stentfix (Experimental)
  Interventions: Device: OTSC Stentfix

INTERVENTIONS:
Device: OTSC Stentfix — Stent placement with fixation of the esophageal stent using OTSC Stentfix.
  Arms: OTSC Stentfix
Procedure: Stent Suturing / Endoscopic Clips — Stent placement with fixation of the esophageal stent using sutures / endoscopic clips.
  Arms: Stent Suturing

SUMMARY:
This study aims to assess the efficacy and rate of stent migration in standard of care esophageal stents that are not fixed, compared to those that are fixed with either standard of care OTSC stentfix or standard of care stent placement with suturing in both benign and malignant esophageal strictures.

ELIGIBILITY:
Inclusion Criteria:

1. The study population will include any adult (18 years +) who will undergo standard of care esophageal stent placement for benign or malignant esophageal strictures as either an inpatient or outpatient at NYULH.
2. The participant is able to consent to stent placements with fixation or without fixation and study procedures, verified by signature on the informed consent form.
3. Willing to comply with all study procedures and be available for the duration of the study.
4. English and Non-English speaking participants.

Exclusion Criteria:

1. Patients who have strictures treated with luman apposing stents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience Stent Migration | Week 48

SECONDARY OUTCOMES:
Total Procedural Time | 120 minutes
  Time it takes to complete standard of care upper endoscopy with standard of care stent placement with or without fixation.
Change in Score on Dysphagia Outcome and Severity Scale (DOSS) | Baseline, Week 48
  DOSS is a simple, easy-to-use, 7-point scale developed to systematically rate the functional severity of dysphagia. The total range of score is 1-7; a lower score indicates more severe symptoms of dysphagia.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Haber, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to sofia.yuen@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.